CLINICAL TRIAL: NCT01857375
Title: A Study of Improved Efficacy, Safety and Compliance to Administer Insulin in Pen vs. Vial and Syringe
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Jeffrey Rothman, Endocrinology, Northwell Health
Other Study IDs: 09-029
Record Dates: First submitted 2013-05-13; First posted 2013-05-20 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes
Keywords: Diabetes - insulin administration
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group receiving insulin via vial/syringe: This group will receive their insulin via vial/syringe
- Insulin Pen: Patients receiving insulin via insulin pen
  Interventions: Device: Insulin Pen Device

INTERVENTIONS:
Device: Insulin Pen Device — Insulin pen was compared to administration of insulin using standard syringes.
  Groups: Insulin Pen

SUMMARY:
This research is to determine the use of insulin pens compared to syringe and vial therapy in adults newly begun on insulin therapy during their hospital stay.

DETAILED DESCRIPTION:
This research is to determine the use of insulin pens compared to syringe and vial therapy in adults newly begun on insulin therapy during their hospital stay. Patients will have no prior experience using insulin or other self-administered injectable medicine. The study will examine which method of administering insulin reduces dosing errors, causes a lower incidence of low blood sugars, increases adherence to therapy and with which method patients are more satisfied.

ELIGIBILITY:
Inclusion Criteria:

* Adult in hospital and diagnosed with diabetes; must have no prior experience using insulin or other self-administered injectable medicine. they must be able to prepare an injection and to self administer the insulin using either a pen device or syringe and vial. They must be willing to monitor their blood sugar three times per day and keep a diary of their sugar measurements and insulin doses.

Exclusion Criteria:

* Previously treated with injectable medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults newly begun on insulin therapy during their hospital stay.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Insulin Dosing Accuracy (in units) | Approximately one year
  Whether the method of administering insulin would: 1) reduce dosing errors as measured by direct observation of patient performance, 2) reduce the risk of hypoglycemia, 3) increase adherence to insulin, 4) improve patient satisfaction.Dosing accuracy was measured by direct observation of subject's performance at follow-up visits.

SECONDARY OUTCOMES:
Reduce the Risk of hypoglycemia (assessed by patient diary) | 3 months
Adherence to prescribed dose of insulin (assess patient diaries and observation of used pens/vials) | 3 months
Patient satisfaction with method of insulin administration measured by questionnaire. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Rothman, MD, Principal Investigator — SIUH